CLINICAL TRIAL: NCT05475769
Title: Nummular Headache Iberian Study on the Treatments and Outcomes in Real-World Setting
Brief Title: NUMITOR Study: Nummular Headache Iberian Study on the Treatments and Outcomes in Real-World Setting
Acronym: NUMITOR
Status: Recruiting | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, David García Azorín, Principal Investigator, Headache Unit, Department of Neurology, Hospital Clínico Universitario de Valladolid
Other Study IDs: PI-GR-21-2394
Record Dates: First submitted 2022-07-15; First posted 2022-07-27 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Headache Disorders, Secondary; Headache Disorders; Central Nervous System Diseases; Brain Diseases; Neurologic Manifestations; Nervous System Diseases; Pain
MeSH Terms: conditions — Headache Disorders, Secondary; Headache Disorders; Central Nervous System Diseases; Brain Diseases; Neurologic Manifestations; Nervous System Diseases; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nummular headache patients: Patients that fulfill the International Classification of Headache Disorders, 3rd edition, for Nummular Headache.
  Interventions: Drug: Clinical evaluation

INTERVENTIONS:
Drug: Clinical evaluation — Patients will receive treatments under the criteria of the responsible physician and the response to these treatments will be prospectively collected.
  Other Names: Patients that under the criteria of the responsible physician receive oral or injectable treatment that are listed in the local Standard of Care

SUMMARY:
The NUMITOR study is an analytical observational study with an multicenter ambisective (retrospective and prospective) cohort design.

DETAILED DESCRIPTION:
This study aims to create a multicenter registry that will increase the knowledge of nummular headache and assess which treatments are more effective and better tolerated. The study population will be patients with nummular headache who, under the opinion of their responsible neurologists, have required or require preventive treatment, in any of its modalities, oral or injectable.

ELIGIBILITY:
Inclusion Criteria:

1. Nummular headache according to the criteria of the International Classification of Headache Disorders, third version (ICHD-3).
2. Nummular headache duration of more than three months.
3. Treatment with a medication with possible preventive drug according to the Clinical Practice Guidelines of the Spanish Society of Neurology21.
4. Age over 18 years.
5. Informed consent signature.

Exclusion Criteria:

1. Diagnosis is better accounted for by any other entity included in the International Classification of Headache Disorders, 3rd version.
2. Serious systemic or psychiatric pathology that makes it difficult to assess the patient.
3. Secondary nummular headache
4. Use of preventive treatment with another indication (e.g., epilepsy, other painful conditions, aesthetic).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be made up of patients with nummular headache who, under the opinion of their responsible neurologists, have required or require preventive treatment, in any of its modalities, oral or injectable.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
50% response 8-12 | Weeks 8-12
  To evaluate the 50% responder rate in patients with NH treated with each preventive drug between weeks 8-12, compared to the baseline situation (month prior to the treatment onset) for each different drug.

SECONDARY OUTCOMES:
50% response 20-24 | Weeks 20-24
  To evaluate the 50% responder rate in the period between weeks 20-24, compared to the baseline situation (month prior to the treatment onset) for each different drug.
30% response 8-12 | Weeks 8-12
  To evaluate the proportion of patients with "partial" response, determined by the 30% response rate, between weeks 8-12, compared to the baseline situation.
30% response 20-24 | Weeks 20-24
  To evaluate the proportion of patients with "partial" response, determined by the 30% response rate, between weeks 20-24, compared to the baseline situation.
75% response 8-12 | Weeks 8-12
  To evaluate the proportion of patients with an "optimal" response, determined by the 75% responder rate, between weeks 8-12, compared to the baseline situation.
75% response 20-24 | Weeks 20-24
  To evaluate the proportion of patients with an "optimal" response, determined by the 75% response rate, between weeks 20-24, compared to the baseline situation.
Adverse events | Weeks 0-24
  To evaluate the frequency and type of treatment-related adverse effects
Adverse events discontinuation | Weeks 0-24
  To evaluate the proportion of patients who discontinue each treatment due to adverse effects.
Response predictors weeks 8-12 | Weeks 0-12
  To calculate which demographic or clinical variables present an odds ratio higher or lower than 1, including the 95% confidence interval, in a logistic regression analysis where the dependent variable is the presence of a 50% responder rate between weeks 8-12.
50% response 8-12 in women | Weeks 0-12
  To evaluate the 50% responder rate in women with NH treated with each preventive drug between weeks 8-12, compared to the baseline situation (month prior to the treatment onset) for each different drug.
Adverse events in women | Weeks 0-24
  To evaluate the frequency and type of treatment-related adverse effects in women
50% response 8-12 in patients older than 65 | Weeks 0-12
  To evaluate the 50% responder rate in patients older than 65 with NH treated with each preventive drug between weeks 8-12, compared to the baseline situation (month prior to the treatment onset) for each different drug.
Adverse events in patients older than 65 | Weeks 0-24
  To evaluate the frequency and type of treatment-related adverse effects in patients older than 65
50% response 8-12 in patients older than 80 | Weeks 0-12
  To evaluate the 50% responder rate in patients older than 80 with NH treated with each preventive drug between weeks 8-12, compared to the baseline situation (month prior to the treatment onset) for each different drug.
Adverse events in patients older than 80 | Weeks 0-24
  To evaluate the frequency and type of treatment-related adverse effects in patients older than 80

CONTACTS AND LOCATIONS:
Overall Officials: David García-Azorín, MD, PhD, Principal Investigator — Hospital Clínico Universitario de Valladolid
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data may be shared upon reasonable request to the principal investigator.

REFERENCES:
- [Background] Pareja JA, Caminero AB, Serra J, Barriga FJ, Baron M, Dobato JL, Vela L, Sanchez del Rio M. Numular headache: a coin-shaped cephalgia. Neurology. 2002 Jun 11;58(11):1678-9. doi: 10.1212/wnl.58.11.1678. PMID 12058099
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Pareja JA, Pareja J, Barriga FJ, Baron M, Dobato JL, Pardo J, Sanchez C, Vela L. Nummular headache: a prospective series of 14 new cases. Headache. 2004 Jun;44(6):611-4. doi: 10.1111/j.1526-4610.2004.446011.x. PMID 15186307
- [Background] Guerrero AL, Martin-Polo J, Gutierrez F, Iglesias F. [Representation of the nummular healdache in general consultation in neurology]. Neurologia. 2008 Sep;23(7):474. No abstract available. Spanish. PMID 18726731
- [Background] Alvaro LC, Garcia JM, Areitio E. Nummular headache: a series with symptomatic and primary cases. Cephalalgia. 2009 Mar;29(3):379-83. doi: 10.1111/j.1468-2982.2008.01722.x. PMID 19220316
- [Background] Porta-Etessam J, Lapena T, Cuadrado ML, Guerrero A, Parejo B. Multifocal nummular headache with trophic changes. Headache. 2010 Nov;50(10):1612-3. doi: 10.1111/j.1526-4610.2010.01773.x. Epub 2010 Oct 12. No abstract available. PMID 21198563
- [Background] Cortijo E, Guerrero-Peral AL, Herrero-Velazquez S, Penas-Martinez ML, Rojo-Martinez E, Mulero P, Fernandez R. [Nummular headache: clinical features and therapeutic experience in a series of 30 new cases]. Rev Neurol. 2011 Jan 16;52(2):72-80. Spanish. PMID 21271546
- [Background] Cortijo E, Guerrero-Peral AL, Herrero-Velazquez S, Penas-Martinez ML, Rojo-Martinez E, Mulero P, Fernandez R. [Nummular headache: shedding light on some concepts. Reply]. Rev Neurol. 2011 Dec 16;53(12):768. No abstract available. Spanish. PMID 22127666
- [Background] Guerrero AL, Cuadrado ML, Garcia-Garcia ME, Cortijo E, Herrero-Velazquez S, Rodriguez O, Mulero P, Porta-Etessam J. Bifocal nummular headache: a series of 6 new cases. Headache. 2011 Jul-Aug;51(7):1161-6. doi: 10.1111/j.1526-4610.2011.01940.x. Epub 2011 Jun 15. PMID 21675970
- [Background] Guerrero AL, Cortijo E, Herrero-Velazquez S, Mulero P, Miranda S, Penas ML, Pedraza MI, Fernandez R. Nummular headache with and without exacerbations: comparative characteristics in a series of 72 patients. Cephalalgia. 2012 Jun;32(8):649-53. doi: 10.1177/0333102412447537. PMID 22711962
- [Background] Mulero P, Matarazzo M, Pedraza MI, Llamas S, Herrero S, Domingo-Santos A, Martinez-Salio A, Guerrero AL. Nummular headache related to exercise or Valsalva maneuver. Clinical characteristics of 3 cases. Headache. 2013 Jul-Aug;53(7):1167-8. doi: 10.1111/head.12133. No abstract available. PMID 23865918
- [Background] Irimia P, Palma JA, Idoate MA, Espana A, Riverol M, Martinez-Vila E. Cephalalgia alopecia or nummular headache with trophic changes? A new case with prolonged follow-up. Headache. 2013 Jun;53(6):994-7. doi: 10.1111/head.12072. Epub 2013 Mar 7. PMID 23469985
- [Background] Herrero-Velazquez S, Guerrero AL, Pedraza MI, Mulero P, Ayllon B, Ruiz-Pinero M, Rojo E, Marco J, Fernandez-Buey N, Cuadrado ML. Nummular headache and epicrania fugax: possible association of epicranias in eight patients. Pain Med. 2013 Mar;14(3):358-61. doi: 10.1111/pme.12022. Epub 2012 Dec 28. PMID 23279627
- [Background] Rodriguez C, Herrero-Velazquez S, Ruiz M, Baron J, Carreres A, Rodriguez-Valencia E, Guerrero AL, Madeleine P, Cuadrado ML, Fernandez-de-Las-Penas C. Pressure pain sensitivity map of multifocal nummular headache: a case report. J Headache Pain. 2015;16:523. doi: 10.1186/s10194-015-0523-7. Epub 2015 Apr 30. PMID 25929432
- [Background] Baron J, Rodriguez C, Ruiz M, Pedraza MI, Guerrero AL, Madeleine P, Cuadrado ML, Fernandez-de-Las-Penas C. Atypical nummular headache or circumscribed migraine: the utility of pressure algometry. Pain Res Manag. 2015 Mar-Apr;20(2):60-2. doi: 10.1155/2015/567072. Epub 2015 Feb 3. PMID 25647287
- [Background] Cuadrado ML, Lopez-Ruiz P, Guerrero AL. Nummular headache: an update and future prospects. Expert Rev Neurother. 2018 Jan;18(1):9-19. doi: 10.1080/14737175.2018.1401925. Epub 2017 Nov 9. PMID 29103335
- [Background] Trigo J, Garcia-Azorin D, Martinez Pias E, Sierra A, Chavarria A, Guerrero AL. Clinical characteristics of nummular headache and differentiation between spontaneous and posttraumatic variant: an observational study. J Headache Pain. 2019 Apr 8;20(1):34. doi: 10.1186/s10194-019-0981-4. PMID 30961529
- [Background] Garcia-Azorin D, Trigo-Lopez J, Sierra A, Blanco-Garcia L, Martinez-Pias E, Martinez B, Talavera B, Guerrero AL. Observational, open-label, non-randomized study on the efficacy of onabotulinumtoxinA in the treatment of nummular headache: The pre-numabot study. Cephalalgia. 2019 Dec;39(14):1818-1826. doi: 10.1177/0333102419863023. Epub 2019 Jul 4. PMID 31272194
- [Background] Clar-de-Alba B, Barriga FJ, Rodriguez-Caravaca G. [Clinical and pathophysiological description of nummular headaches: a case series]. Rev Neurol. 2020 Mar 1;70(5):171-178. doi: 10.33588/rn.7005.2019152. Spanish. PMID 32100277
- [Background] Patel UK, Saleem S, Anwar A, Malik P, Chauhan B, Kapoor A, Arumaithurai K, Kavi T. Characteristics and treatment effectiveness of the nummular headache: a systematic review and analysis of 110 cases. BMJ Neurol Open. 2020 Mar 12;2(1):e000049. doi: 10.1136/bmjno-2020-000049. eCollection 2020. PMID 33681785
- [Background] Tassorelli C, Diener HC, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of preventive treatment of chronic migraine in adults. Cephalalgia. 2018 Apr;38(5):815-832. doi: 10.1177/0333102418758283. Epub 2018 Mar 4. PMID 29504482
- [Background] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Background] Chavarria-Miranda A, Guerrero AL, Talavera B, Martinez-Pias E, Trigo-Lopez J, Sierra A, Garcia-Azorin D. Linear Headache: A Novel Entity or a Variant of Nummular Headache? Clinical Characteristics and Treatment Response in a Series of 16 Patients. Pain Med. 2021 May 21;22(5):1158-1166. doi: 10.1093/pm/pnaa436. PMID 33723599
- [Background] Garcia-Iglesias C, Martinez-Badillo C, Garcia-Azorin D, Trigo-Lopez J, Martinez-Pias E, Guerrero-Peral AL. Secondary Nummular Headache: A New Case Series and Review of the Literature. Pain Med. 2021 Nov 26;22(11):2718-2727. doi: 10.1093/pm/pnab174. PMID 34022054

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-07-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT05475769/SAP_001.pdf